CLINICAL TRIAL: NCT01793805
Title: NSABP Patient Registry and Biospecimen Profiling Repository
Status: Completed | Type: Observational
Sponsor: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Other Study IDs: NSABP MPR-1
Record Dates: First submitted 2013-02-11; First posted 2013-02-18 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tissue blocks from the primary tumor site and an uninvolved margin of resection (normal tissue).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic Colorectal Cancer Patients

SUMMARY:
This is a study to collect and analyze tissue specimens from metastatic colorectal cancer (mCRC) patients for the development of a molecularly profiled tissue repository for the primary purpose of maintaining a patient registry for future clinical trials based on the molecular profile of the tumors. The main purpose of testing these tissue specimens is to identify genetic alterations or biomarkers associated with colorectal cancer such that if new agent(s) become available, particularly those that target these genetic alterations/biomarkers, participants may be offered the opportunity to take part in a National Surgical Adjuvant Breast and Bowel Project (NSABP) treatment protocol.

DETAILED DESCRIPTION:
Tissue blocks from the primary tumor site and an uninvolved margin of resection (normal tissue) from consenting patients will be submitted and stored at the NSABP Division of Pathology, in the NSABP Biospecimen Profiling Repository. Tissue specimens will be used to profile molecular characteristics, including actionable mutations most commonly identified in colorectal cancer. Specimens may be further interrogated by other methods to discover additional mechanisms and targetable genetic alterations that may predict sensitivity or resistance to drug therapies.

The repository will be populated, maintained, and analyzed through continuous patient recruitment. Patient tumor specimens will be interrogated to characterize an individual's molecular profile. At a future date for discovery purposes, the normal tissue may be profiled for comparison with the profile of the tumor tissue. NSABP will hold a database with molecular profiles and relevant patient information. As agents become available for clinical study, particularly those matching specified profiles, the treating physician will be contacted so that the patient may be offered participation in that trial via a separate consent process. Each NSABP trial will have a defined molecular profile for entry which will be specific to the agent(s) under study. The MPR-1 patient registry and tissue repository and all treatment protocols associated with MPR-1 are being developed as part of the NSABP Oncology-Genome Assessment Guided Medicine (N-GAMe) Program.

This registry and repository platform uses a translational science approach for more personalized therapy for patients with mCRC. This analysis provides an individual molecular profile in an attempt to direct each patient's treatment based on the pattern of genetic alterations. These efforts also may aid in the discovery of with or without new gene targets for future drug development.

Approximately 1000-2000 tumor (with or without) normal tissue specimens from living mCRC patients will be collected, stored, and analyzed as part of this biospecimen repository. It is anticipated that 200-400 participants will be registered within the first year.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a diagnosis of metastatic colorectal adenocarcinoma.
* Representative formalin-fixed paraffin-embedded (FFPE) tissue blocks from the primary colorectal tumor surgery with corresponding pathology report must be available for release by the local pathology department (an adequate amount of tumor tissue is required for analysis). If available for release, a separate FFPE tissue block from an uninvolved margin of colorectal resection (normal tissue) is also requested.
* The patient must have a life-expectancy of greater than or equal to 6 months.

Exclusion Criteria:

* History of non-CRC malignancy unless the patient is considered by the physician to be disease-free and at low risk for recurrence.
* Known comorbid medical conditions that would preclude investigational treatment (e.g., active hepatitis B or C; symptomatic cardiac disease; renal insufficiency; bone marrow impairment).
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude investigational treatment.
* Colonoscopy biopsies or diagnostic core biopsy procedures without surgery or resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic colorectal cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 3232 (Actual)
Dates: Start 2013-02; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
To characterize common genetic/molecular profiles associated with colorectal cancer (CRC) | From start of study through study completion at approximately 6 months
  This is a living registry with no end date provided continued funding.

SECONDARY OUTCOMES:
To identify subpopulations of registry patients on the basis of their molecular profiles that may be eligible for participation in available NSABP clinical trials involving novel agents | From start of study through study completion at approximately 6 months
To conduct further analysis of tumor samples for the discovery of new potential targets and mechanisms of drug resistance | From start of study through study completion at approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (46):
- United States (46):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-San Diego, San Diego, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - University of Florida, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Kootenai Health Cancer Services, Post Falls, Idaho
  - Decatur Memorial Hospital, Decatur, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medstar Franklin Square Medical Center, Weinberg Cancer Institute, Baltimore, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - CCOP, Kalamazoo, MI, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - CCOP - Cone Health Cancer Center, Greensboro, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - CCOP Forsyth Memorial Hospital, Winston-Salem, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital/Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Cancer Centers of the Carolinas (International), Greenville, South Carolina
  - CCOP - Sanford Research, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - MBCCOP, Virginia Commonwealth University, Richmond, Virginia
  - CCOP, St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP, Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Health Care, Milwaukee, Wisconsin